CLINICAL TRIAL: NCT05084391
Title: Phase I/II Randomized Study of Stereotactic Ablative Radiotherapy (SABR) Versus Standard of Care for Refractory Structural Cardiac Arrhythmias (SABR-HEART)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0538; NCI-2021-10672 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2021-09-03; First posted 2021-10-19 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Arrhythmia; Cardiac; Ventricular Tachyarrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Phase I: (Experimental): Phase I there will be up to 15 patients treated with SABR and followed for 6 months post-treatment to ensure no significant acute grade 3 or 4 toxicity from SABR treatment.
  Interventions: Device: stereotactic ablative radiotherapy (SABR); Other: Standard of Treatment
- Phase II (Experimental): Phase II portion with 25 patients in each arm assigned to SABR or current practice (standard of care)
  Interventions: Device: stereotactic ablative radiotherapy (SABR); Other: Standard of Treatment

INTERVENTIONS:
Device: stereotactic ablative radiotherapy (SABR) — is safe for treating heart arrhythmias (irregular heartbeat
Other: Standard of Treatment — Standard of care

SUMMARY:
Phase I: For the Phase I portion, there will be up to 15 patients treated with SABR and followed for 6 months post-treatment to ensure no significant acute grade 3 or 4 toxicity from SABR treatment. Efficacy as defined below will also be assessed. Following this Phase I lead-in, results will be presented to the FDA for review. Only upon favorable analysis by the FDA committee, and with written explicit permission, will the Phase II randomized portion ensue. This is to act as a safety and efficacy safeguard and has is addressed more thoroughly in the Statistical Analysis Plan of this protocol.

Phase II: A 1:1 randomized Phase II portion with 25 patients in each arm assigned to SABR or current practice (standard of care; Figure 3). Standard of care is defined as nationally recognized appropriate next treatment strategies for medical and catheter-ablation refractory structural cardiac VT that is assessed and judged appropriate for the patient by his/her treating cardiologist. This includes repeat catheter ablation (intravascular and/or epicardial catheter ablation), placement of left-ventricular assist device (LVAD), heart transplant, or further medical management (e.g. antiarrhythmic drug modulation/continuation). Randomization will be performed through the Clinical Trial Conduct (CTC) website.

DETAILED DESCRIPTION:
Primary Objectives Phase I:

-Assess acute toxicity and efficacy with SABR in treating refractory structural cardiac ventricular tachyarrhythmias (VT). Ensure safety and treatment efficacy.

Primary Objectives Phase II:

* Investigate overall toxicity with SABR compared to next best management practices (standard of care) in treating refractory structural cardiac ventricular tachyarrhythmias (VT).
* Investigate VT episode reduction with SABR compared to standard of care to evaluate effectiveness and potential superiority of SABR to current day options.

Primary Objectives Phase I:

1. Assess acute toxicity and efficacy with SABR in treating refractory structural cardiac ventricular tachyarrhythmias (VT). Ensure safety and treatment efficacy.

Primary Objectives Phase II:

1. Investigate overall toxicity with SABR compared to next best management practices (standard of care) in treating refractory structural cardiac ventricular tachyarrhythmias (VT).
2. Investigate VT episode reduction with SABR compared to standard of care to evaluate effectiveness and potential superiority of SABR to current day options.

Secondary Objectives

The following endpoints will be analyzed retrospectively based on prospectively collected (event-free survival endpoints) and at the specified time points (e.g. QOL questionnaire). Participation in QOL assessment and bio specimen collection for secondary endpoints is completely voluntary and not mandated by the trial.

1. 6-month and 1-year overall survival (OS) of SABR compared to standard of care.
2. Quality of life (QOL) with SABR compared to standard of care (baseline and at 6 months after randomization).
3. Hospitalization-free survival with SABR compared to standard of care (evaluated at 1-year).
4. Cost-effectiveness analysis with SABR compared to standard of care (evaluated at 1-year).
5. Freedom-from Antiarrhythmic medications with SABR compared to standard of care (evaluated at 1-year).
6. Freedom-from Electrical Storm with SABR compared to standard of care (evaluated at 1-year).
7. Treatment-free Survival with SABR compared to standard of care (evaluated at 1-year).
8. Event-free Survival with SABR compared to standard of care (evaluated at 1-year).
9. Long term (>1year) toxicity with SABR compared to standard of care (evaluated at 1-year).
10. Ejection fraction improvement with SABR compared to standard of care (evaluated at 1-year).
11. Transplant/LVAD-free survival with SABR compared to standard of care (evaluated at 1-year).
12. Number, type, and treatment success and cycle length of ICD-treated VTs with SABR compared to standard of care (evaluated at 1-year).
13. Parameters obtained from cardiac imaging, and/or serum markers will be associated with frequency of survival, response to treatment, and toxicity at regular time intervals using cardiac ECHO, MRI, CT imaging, ICD interrogation, and/or serum/blood work studies for prognostic/predictive biomarker and radiomic identification.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG 0-2
2. Age 18 years or older
3. Diagnosis of recurrent sustained monomorphic VT (MMVT) in the setting of structural heart disease.
4. ICD placement and at least two (2) episodes of recurrencerecurrent sustained MMVT that are terminated by anti-tachycardia pacing (ATP) or ICD shocks confirmed by device interrogation in the preceding 3 months, since the last VT ablation procedure in subjected who have failed catheter ablation.
5. Failed at least 1 anti-arrhythmic medication (not including beta-blockers) as evidenced by persistent VT (including amiodarone and/or sotalol)
6. At least 1 attempted catheter ablation procedure with voltage and/or activation 3D mapping. For patients with ischemic cardiomyopathy this would include failure of at least one endocardial ablation performed at an experienced center. For patients with non-ischemic cardiomyopathy, both endocardial and epicardial ablation should have been attempted unless epicardial ablation/mapping is not feasible (e.g. patient tolerance, deemed futile by EP, prior cardiac surgery).
7. Patients are eligible regardless of past or present oncologic history (however, please refer to exclusion criterion #1 below, regarding life-expectancy of at least 12 months in the absence of VT)

Exclusion Criteria:

1. Unlikely to live at least 12 months in the absence of VT, as assessed by physicians
2. Heart failure dependent on ionotropes
3. Left ventricular assist device
4. Polymorphic VT
5. Ventricular fibrillation
6. 5 or more VT morphologies during stimulation testing suggestive of more than one arrhythmogenic substrate
7. Prior radiation treatment to the chest for any reason
8. Last invasive catheter ablation attempt <2 weeks
9. Lack of ICD data in preceding 3 months
10. Unable/unwilling to provide informed consent
11. Idiopathic VT
12. Women who are pregnant
13. Heart transplant
14. Active ischemia or other reversible causes of VT
15. Active non-cardiovascular illness or systemic infection
16. Cardiogenic shock
17. Presence of incessant VT that is hemodynamically unstable
18. Acute heart failure exacerbation
19. Revascularization in the past 30 days
20. Left ventricular ejection fraction <15%
21. Scar tissue exceeding 80cc in volume planning treatment volume (PTV) ≥300cc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
The overall toxicity as assessed using CTCAE v4.0 will be used with SABR compared to next best management practices (standard of care) in treating refractory structural cardiac ventricular tachyarrhythmias (VT). | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joe Chang, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org